CLINICAL TRIAL: NCT04842383
Title: Androgenetic Alopecia Treatment Using Varin and Cannabidiol-rich Topical Hemp Oil - A Case Series
Brief Title: Androgenetic Alopecia Treatment Using Varin and Cannabidiol Rich Topical Hemp Oil: A Case Series
Acronym: Hair Regrowth
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gregory L Smith, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Gregory L Smith, MD, MPH, Primary Investigator, Medical Life Care Planners, LLC
Organization: Medical Life Care Planners, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alopecia Treated with Hemp oil
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — hempseed oil; cannabidivarin; peppermint oil

STUDY DESIGN:
Intervention Model Description: 40 subjects will be randomly assigned into two treatment groups, 500mg of cannabinoids per ounce and 1000mg of cannabinoids per ounce. The change in hair follicle numbers will be compared statistically between the two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants in the study and the outcomes assessor on day 0 and day 180 will be prevented from having knowledge of which of the two strengths of cannabinoid topicals were used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Half strength Hemp Oil Preparation (Active Comparator): The topical preparation contains only 500mg of cannabinoids per ounce. The other ingredients are the same in both arms.
  Interventions: Drug: Hemp Oil
- Full strength Hemp Oil Preparation (Active Comparator): The topical preparation contains 1000mg of cannabinoids per ounce. The other ingredients are the same in both arms.
  Interventions: Drug: Hemp Oil

INTERVENTIONS:
Drug: Hemp Oil — Hemp oil extract rich in varins (THCV and CBDV) as well as cannabidiol (CBD) in combination with 3% peppermint oil extract
  Other Names: THCV, tetrahydrocannabivarin, CBDV, cannabidivarin, peppermint oil

SUMMARY:
This is a case series of adult, male and female subjects with androgenetic alopecia (male pattern baldness). A topical hemp oil that is rich in varins (THCV and CBDV) and cannabidiol (CBD) is being used daily for six months to stimulate hair regrowth using Endocannabinoid System (ECS) receptors that are found on hair follicles.

DETAILED DESCRIPTION:
The study is a case series of adults (males and females) presenting to a "Hair and Scalp" center in Clearwater, Florida. Subjects diagnosed with androgenetic alopecia (AGA - male pattern baldness) and who were not currently using minoxidil or finasteride, were offered the opportunity to receive a topical hemp-oil extract that is high in varins (tetrahydrocannabivarin, (THCV) cannabidivarin (CBDV)) as well as cannabidiol (CBD). The topical also contains 3% peppermint oil. The subjects were given the topical free of charge. Subjects were randomly assigned to one of two doses, 500mg of hemp oil per dispenser or 1000mg per dispenser. Each dispenser lasted approximately one month, so they used either 1.7mg or 3.4 mg of hemp extract per day.

Forty subjects withAGA with Norwood-Hamilton Classification score of 3V or higher will be selected randomly. The predefined endpoints were hair counts obtained in a defined, representative area of scalp hair loss using a small tattoo to confirm the location of measuring hair loss. The primary investigator will make a clinical assessment of hair growth.

The subjects gave their written informed consent for this six-month trial. The study adhered to the Helsinki guidelines and was institutionally approved. None of the subjects were currently using minoxidil or finasteride. No other hair loss treatments were used during the six months of the research.

The subjects were randomly assigned to using a dropper bottle or spray can with a nozzle to apply the extract. Subjects are advised to apply a thin layer once each morning to the areas of baldness. The hemp oil extract with peppermint was independently analyzed The hemp oil was infused into a lanolin base lotion and natural Emu oil carrier. Each container (dropper bottle or spray can) contained one ounce of the extract. Each container is expected to last approximately one month. The subjects were advised that they could use blow dryers, conditioners, and other hair preparations. The hemp extract was replaced as needed throughout the six-month trial.

A hair count of the greatest area of alopecia was carried out before treatment was started and again after six months of treatment. To facilitate consistent hair count analysis, a small permanent black tattoo, approximately 1mm in diameter, was applied to each subject's head at the area of greatest alopecia. The nonvellus hairs within the 1 cm2 cutout were pulled through the opening with a surgical skin hook and a hair count was taken using a Bodelin ProScope with 50x magnification.

Statistical analysis was done comparing the number of nonvellus hairs in the 1cm2 cutout before and after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older

Physician-diagnosed androgenetic alopecia (AGA) with Norwood-Hamilton Classification score of 3V or higher.

Not currently using minoxidil or finasteride.

Agree to complete six months of the study.

Agreed to not use other hair loss treatments, including minoxidil and/or finasteride during the six months of the study.

Agrees to and signs Informed Consent Form.

Exclusion Criteria:

Inability to meet the 'Inclusion Criteria' above.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-10-04 (Estimated); Study Completion 2021-10-04 (Estimated)

PRIMARY OUTCOMES:
Change in nonvellus hair count in 1cm2 area of the bald scalp | six months
  Change in nonvellus hair count in standard area of the bald scalp

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Smith, MD, Principal Investigator — Medical Life Care Planners, LLC
Locations (1):
- Hair and Scalp Clinic, Clearwater, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baswan SM, Klosner AE, Glynn K, Rajgopal A, Malik K, Yim S, Stern N. Therapeutic Potential of Cannabidiol (CBD) for Skin Health and Disorders. Clin Cosmet Investig Dermatol. 2020 Dec 8;13:927-942. doi: 10.2147/CCID.S286411. eCollection 2020. PMID 33335413
- [Background] Telek A, Biro T, Bodo E, Toth BI, Borbiro I, Kunos G, Paus R. Inhibition of human hair follicle growth by endo- and exocannabinoids. FASEB J. 2007 Nov;21(13):3534-41. doi: 10.1096/fj.06-7689com. Epub 2007 Jun 12. PMID 17567570
- [Background] Sugawara K, Zakany N, Tiede S, Purba T, Harries M, Tsuruta D, Biro T, Paus R. Human epithelial stem cell survival within their niche requires "tonic" cannabinoid receptor 1-signalling-Lessons from the hair follicle. Exp Dermatol. 2021 Apr;30(4):479-493. doi: 10.1111/exd.14294. Epub 2021 Feb 26. PMID 33523535
- [Background] Smith GL, Satino J. Hair Regrowth with Cannabidiol (CBD)-rich Hemp Extract - A Case Series. Cannabis. 2021 Apr 22;4(1):53-59. doi: 10.26828/cannabis/2021.01.003. eCollection 2021. PMID 37287996